CLINICAL TRIAL: NCT02780336
Title: Diagnostic and Rating Tools for Blepharospasm
Brief Title: Blepharospasm Tools
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Benign Essential Blepharospasm Research Foundation (Other)
Responsible Party: Principal Investigator, Hyder A. Jinnah, MD, PhD, Principal Investigator, Emory University
Other Study IDs: IRB00087047; U54TR001456 (NIH)
Record Dates: First submitted 2016-05-18; First posted 2016-05-23 (Estimated); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Blepharospasm; Dystonia; Other Eye and Face Disorders
MeSH Terms: conditions — Blepharospasm; Dystonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Blepharospasm (BL): Participants in this group should be diagnosed with blepharospasm, but may have dystonia in other body parts as well.
  Interventions: Other: No intervention.
- Disease Control Group: Participants in this group should be diagnosed with a disorder affecting their eyes or face, such as hemifacial spasm, facial tics, or apraxia.
  Interventions: Other: No intervention.
- Normal Control Group: Participants in this group should not have any neurologic problems or other disorders affecting patients eyes or face.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — Participants will complete questionnaires and interviews as well as have a neurological exam that will be video recorded. For this exam they will do simple movements (like looking at the camera, squeezing your eyes closed, moving your head, and writing).

SUMMARY:
The aim of this study is to develop new rating scales to help diagnose and measure the severity of blepharospasm. This is a condition involving a lot of blinking and spasms of eye closure that people can't control. This study will also test some video software to see if it can help diagnose people or tell the severity of disease using only a video recording of an exam. There is an additional plan to create an educational video to teach others the proper use of the scale and video software.

DETAILED DESCRIPTION:
Blepharospasm is a chronic disorder characterized by too many contractions in the muscles around the eye and nearby facial muscles, leading to involuntary eye closure. This study involves a comprehensive evaluation for patients with blepharospasm, other eye and face disorders, and people without any neurologic or eye or face disorders. It addresses abnormal movements of the muscles around the eye, pain in those muscles, psychological accompaniments, and impact on regular daily life. The evaluation for each participant will be done on a single visit, and it may take up to 1.5 hours to complete. Each participant in this study will be asked to do the following:

* Provide a copy of medical records and provide a medical history relating to the diagnosis of blepharospasm.
* Have an examination by a neurologist or ophthalmologist to reveal the features and extent of dystonia or other eye and face disorders. The examination will be video recorded so it can be reviewed later by different experts.
* Complete some questionnaires about quality of life and psychiatric well being

The doctors will also complete various scales and questionnaires based on the participant's study visit.

ELIGIBILITY:
BLEPHAROSPASM (BL) GROUP

Inclusion Criteria:

* Diagnosed with Focal, Multifocal or Segmental Isolated Dystonia with Onset in Adulthood, must include blepharospasm.
* Sufficiently symptomatic at recruitment to ensure that (eye) problems are evident to evaluators.
* Has ability to provide informed consent and follow study directions.

Exclusion Criteria:

* Evidence of a secondary cause for dystonia as defined as blepharospasm caused by drug exposure, parkinsonism, or stroke.
* Suspected psychogenic movement or eye disorders.
* Has had surgical intervention for blepharospasm or eye problems that may confound interpretations, such as orbital myectomy, blepharoplasty, or deep brain stimulation surgery.
* Is being treated with dopamine receptor antagonists.
* Received BTX injection/botulinum toxin less than 10 weeks prior to study visit.
* Taking any concomitant medications that haven't been at stable doses for at least 1 month prior to study enrollment.
* Has significant medical or neurological conditions that preclude completing the video protocol and questionnaires.
* Has significant physical or other condition that would confound diagnosis or evaluation.

DISEASE CONTROL GROUP:

Inclusion Criteria:

* Diagnosed with a facial or eye disorder that can be confused with blepharospasm, including, but not limited to, hemifacial spasm, facial tics, psychogenic facial disorders, apraxia, and ptosis due to weakness. It is permissible for these problems to be part of Bell's palsy, myasthenia gravis, or Progressive Supranuclear Palsy (PSP).
* Has no significant dystonia in any body part.
* Sufficiently symptomatic at recruitment to ensure that (eye) problems are evident to evaluators.
* Has ability to provide informed consent and follow study directions.

Exclusion Criteria:

* Significant dystonia.
* Evidence of secondary blepharospasm as defined as blepharospasm caused by drug exposure or stroke.
* Received BTX injection/botulinum toxin less than 10 weeks prior to study visit.
* Taking any concomitant medications that haven't been at stable doses for at least 1 month prior to study enrollment.
* Unable to provide informed consent and follow study directions.
* Has significant medical or neurological conditions that preclude completing the video protocol and questionnaires.
* Has significant physical or other condition that would confound diagnosis or evaluation.

NORMAL CONTROL GROUP:

Inclusion Criteria:

* Has no facial or eye problem and no other neurological complaints.

Exclusion Criteria:

* Has facial or eye problem or other neurological complaints.
* Taking any concomitant medications that haven't been at stable doses for at least 1 month prior to study enrollment.
* Unable to provide informed consent and follow study directions.
* Has significant medical or neurological conditions that preclude completing the video protocol and questionnaires.
* Has significant physical or other condition that would confound diagnosis or evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators hope to recruit 200 participants with blepharospasm, about 150 with other eye and face disorders, and 50 with no neurologic, eye or face disorder.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2016-08; Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Blepharospasm Diagnostic Rating Scale (BDRS) | Day 1
  The ratings for the BDRS will be examined for internal consistency by pair-wise correlations among all items in the scale in all combinations of possible pairs.
Blepharospasm Severity Rating Scale (BSRS) | Day 1
  The ratings for the BSRS will be examined for internal consistency by pair-wise correlations among all items in the scale in all combinations of possible pairs.
Blepharospasm Screening Questions - Motor (BSQ-M) | Day 1
Blepharospasm Screening Questions - Psych (BSQ-P) | Day 1
  Concurrent validity for the BSQ-P will be assessed using correlations between the responses to the questionnaire and data from the corresponding scales included in the concurrent validity packet (BDI-II, HADS, LSAS and PHQ-9).
Blepharospasm Disability Index (BSDI) | Day 1

SECONDARY OUTCOMES:
Craniocervical Dystonia Questionnaire (CDQ-24) | Day 1
Eye Symptoms in Blepharospasm | Day 1
Jankovic Rating Scale (JRS) | Day 1
Oromandibular Dystonia Questionnaire (OMDQ-25) | Day 1
Obsessive Compulsive Inventory-Revised Edition (OCI-R) | Day 1
Global Dystonia Rating Scale (GDRS) | Day 1
Fahn-Marsden Dystonia Scale (FM) | Day 1
Beck Depression Inventory II (BDI-II) | Day 1
  Concurrent validity for the BSQ-P will be assessed using correlations between the responses to the questionnaire and data from the corresponding scales included in the concurrent validity packet (BDI-II, HADS, LSAS and PHQ-9).
Patient Health Questionnaire 9 (PHQ-9) | Day 1
  Concurrent validity for the BSQ-P will be assessed using correlations between the responses to the questionnaire and data from the corresponding scales included in the concurrent validity packet (BDI-II, HADS, LSAS and PHQ-9).
Hospital Anxiety and Depression Scale (HADS) | Day 1
  Concurrent validity for the BSQ-P will be assessed using correlations between the responses to the questionnaire and data from the corresponding scales included in the concurrent validity packet (BDI-II, HADS, LSAS and PHQ-9).
Liebowitz Social Anxiety Scale (LSAS) | Day 1
  Concurrent validity for the BSQ-P will be assessed using correlations between the responses to the questionnaire and data from the corresponding scales included in the concurrent validity packet (BDI-II, HADS, LSAS and PHQ-9).
Short Form Health Survey-36 Quality of Life Scale (SF-36) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: H. A. Jinnah, MD, PhD, Principal Investigator — Emory University
Locations (11):
- United States (7):
  - University of Colorado Denver, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health, Bethesda, Maryland
  - Washington University in St. Louis, St Louis, Missouri
  - Baylor College of Medicine, Houston, Texas
- Toronto Western Hospital, Toronto, Ontario, Canada
- University Hospital of Schleswig-Holstein, Lübeck, Germany
- Italy (2):
  - University of Bari, Bari
  - University of Rome, Rome

REFERENCES:
- See also: Study description on Dystonia Coalition website — http://www.rarediseasesnetwork.org/cms/dystonia/Get-Involved/Research-Studies/6304